CLINICAL TRIAL: NCT03996252
Title: Combination Calcipotriene 0.005% Foam and Fluorouracil 5% Cream for the Treatment of Actinic Keratoses on the Scalp
Brief Title: Combination Topical Therapy for Treatment of Scalp Actinic Keratoses
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: The study team was not able to start the study and they never completed the IRB submission, so the study was terminated.
Sponsor: Tulane University (Other)
Collaborators: Mayne Pharma International Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 052090
Record Dates: First submitted 2019-06-20; First posted 2019-06-24 (Actual); Last update posted 2020-12-07 (Actual); Status verified 2020-12

CONDITIONS: Actinic Keratoses
MeSH Terms: conditions — Keratosis, Actinic | interventions — calcipotriene; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Combination treatment arm (Experimental): Combination of calcipotriene 0.005% foam (Sorilux) and Fluorouracil Cream, 5% USP (generic) applied for four consecutive nights for the treatment of scalp actinic keratoses.
  Interventions: Drug: Calcipotriene 0.005% Foam; Drug: Efudex 5% Topical Cream

INTERVENTIONS:
Drug: Calcipotriene 0.005% Foam — Application of calcipotriene foam in conjunction with generic efudex cream to the scalp for four consecutive nights for the treatment of scalp actinic keratoses
  Other Names: Calcipotriene; Sorilux
Drug: Efudex 5% Topical Cream — Application of generic efudex cream in conjunction with calcipotriene foam to the scalp for four consecutive nights for the treatment of scalp actinic keratoses
  Other Names: Efudex; 5-fluorouracil 5% cream

SUMMARY:
The aim of this study is to determine the effectiveness of combination calcipotriene 0.005% foam and 5% fluorouracil cream for the treatment of actinic keratoses on the scalp. The data obtained will be compared with the current standard of care, monotherapy with 5% fluorouracil cream. A recent randomized, double-blind clinical trial (NCT02019355) compared 0.005% calcipotriol ointment and fluorouracil 5% cream with Vaseline plus fluorouracil 5% cream for a 4-day treatment of actinic keratoses on the face, scalp and upper extremities. They found that calcipotriol plus 5-FU versus Vaseline plus fluorouracil 5% cream led to an 87.8% versus 26.3% mean reduction in the mean number of actinic keratoses. Our study will independently assess the effectiveness of combination treatment (calcipotriene 0.005% foam and fluorouracil 5% cream) on scalp actinic keratoses in a case series of up to 15 eligible participants. Participants will complete a 4-night application of combination treatment with follow-up immediately after and 8 weeks later.

ELIGIBILITY:
Inclusion Criteria:

* Age of at least 40 years.
* Presence of four to fifteen clinically typical, visible, and discrete actinic keratoses in 25 cm2 on the scalp.
* Ability and willingness of the patient to participate in the study (Informed consent is obtained)

Exclusion Criteria:

* Treatment area is within 5 cm of an incompletely healed wound or a suspected basal-cell or squamous-cell carcinoma
* Treatment area contains hypertrophic/hyperkeratotic lesions, cutaneous horns, or lesions that had not responded to repeated cryotherapy
* Recent (within a month) use of medications that could interfere with evaluation of the treatment area (e.g., topical medications, artificial tanners, immunosuppressive medications, immunomodulating agents, cytotoxic drugs, ultraviolet B phototherapy, other therapies for actinic keratoses, or oral retinoids)
* Premenopausal Women (to avoid any risk of pregnancy)
* History of hypercalcemia or clinical evidence of vitamin D toxicity (avoidance of calcipotriene toxicity).

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-06-08 (Actual)

PRIMARY OUTCOMES:
Percentage of change in the number of scalp actinic keratoses from baseline | 8 weeks
  Determine the efficacy of calcipotriene 0.005% foam and 5-fluorouracil 5% cream for the treatment of scalp actinic keratoses following 4 nights of combination treatment. The outcome of interest is percentage change from baseline number of actinic keratoses in the target treatment area on scalp at 8 weeks after treatment.

SECONDARY OUTCOMES:
Complete and partial (>75%) clearance of actinic keratoses | 8 weeks
  To determine complete and partial (>75%) clearance of actinic keratoses at 8 weeks after treatment.
Composite score of erythema, itching and skin pain after topical of calcipotriene 0.005% foam and 5-fluorouracil 5% cream application for four consecutive nights to scalp actinic keratoses. | 4 days
  To determine the composite scores of erythema, itching and pain (determined using standardized scales) following topical application of of calcipotriene 0.005% foam and 5-fluorouracil 5% cream application for four consecutive nights to scalp actinic keratoses.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Powell, MD, Principal Investigator — Tulane Department of Dermatology
Locations (1):
- Tulane University Medical Center, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cunningham TJ, Tabacchi M, Eliane JP, Tuchayi SM, Manivasagam S, Mirzaalian H, Turkoz A, Kopan R, Schaffer A, Saavedra AP, Wallendorf M, Cornelius LA, Demehri S. Randomized trial of calcipotriol combined with 5-fluorouracil for skin cancer precursor immunotherapy. J Clin Invest. 2017 Jan 3;127(1):106-116. doi: 10.1172/JCI89820. Epub 2016 Nov 21. PMID 27869649